CLINICAL TRIAL: NCT06699927
Title: A Feasibility Study of Working Memory Training for People Aging with HIV
Brief Title: Working Memory Training for People Aging with HIV
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NU-20241107
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Cognitive Change

STUDY DESIGN:
Intervention Model Description: A randomized crossover trial will be conducted and participants will be randomly assigned to 1 of 2 conditions: Condition 1 consists of training type 1 followed by training type 2, whereas Condition 2 consists of training type 2 followed by training type 1. They will be assigned to Non-Gamified Span training and Gamified Span training.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-gamified First (Active Comparator): Training type 1 will be administered in the first part of the crossover trial and Training type 2 will be administered in the second part of the trial. Each training part consists of 20 twenty-minute long sessions with the recommended frequency of 2 sessions per work day. Thus each training part can be completed in 10 work days (2 weeks).
  Interventions: Behavioral: Span
- Gamified First (Active Comparator): Training type 2 will be administered in the first part of the crossover trial and Training type 1 will be administered in the second part of the trial. Each training part consists of 20 twenty-minute long sessions with the recommended frequency of 2 sessions per work day. Thus each training part can be completed in 10 work days (2 weeks).
  Interventions: Behavioral: Span

INTERVENTIONS:
Behavioral: Span — The training program is a personal device-based adaptive version of a visual working memory span task, either devoid of game elements or embedded in a gamified platform game

SUMMARY:
The present study investigates the feasibility of working memory training in people aging with HIV (PAWHIV). In a cross-over design this stage 1 feasibility trial, will evaluate acceptability, and estimate possible effect sizes related to working memory training by examining potential differential effects in PAWHIV and those aging without HIV. This project highlights the importance of tailored cognitive assessments and interventions, engaging with underrepresented communities to enhance inclusivity in cognitive health research.

DETAILED DESCRIPTION:
In a randomized controlled trial (RCT) with a 3x2 design (pre-test, post-test, follow-up; PAWHIV, people aging without HIV), we will evaluate feasibility of implementing working memory-based interventions in PAWHIV. This study will examine the differential effects of WM training between PAWHIV and aging adults without HIV, providing insight into specific cognitive challenges in PAWHIV that may influence the efficacy of cognitive training interventions. The results of this trial will be instrumental in developing targeted, evidence-based interventions that promote cognitive health for PAWHIV and contribute to the broader understanding of cognitive aging in vulnerable populations.

Relying on an extended battery of cognitive assessments, we will test different multivariate models to best capture the unique cognitive profiles of PAWHIV and how they compare with people aging without HIV. This analytical framework will allow us to gain insight into and better addressing the needs of the PAWHIV community

The cross-over trial will obtain within-subject comparisons of training with enriched (game-like) versions of working memory training tasks compared to basic (non-gamified) versions of these tasks. Participants are assigned to Non-Gamified Span training and Gamified Span training for a total of 50 sessions per participant: the first few sessions consist of completing questionnaires and computerized cognitive assessments (pre-test). Participants then complete 20 sessions of working memory training. After a mid-test, they complete 20 sessions of a different type of working memory training. Post-test is administered upon training completion, and at least a month later, participants complete 3 follow-up sessions.

ELIGIBILITY:
Inclusion Criteria:

* 50-85 years of age
* Able to understand and speak English and follow study procedures
* Does not have a psychological or neurological condition that would prevent being able to give consent to participate
* Not currently involved in any other cognitive or memory training studies

Exclusion Criteria:

* Formal diagnosis of dementia or other neurological disease, including Mild cognitive impairment.
* A final total score below 17 on Montreal Cognitive Assessment - Blind (telephone) version.
* Score of 10 or more on the Generalized Anxiety Questionnaire (GAD7; Spitzer et al., 2006, Archives of Internal Medicine), indicating presence of moderate or severe anxiety
* Score of 9 or more on Geriatric depression scale (GDS15; Yesavage et al., 1982) indicating presence of moderate or severe depression
* Abnormal visual acuity prohibitive of tablet-based training.
* Physical handicap (motor or perceptual) that would impede training procedures.
* Medical illness requiring treatment and/or significant absences during the study timeline.
* Current evidence or 2-yr history of seizures, focal brain lesion, or head injury with loss of consciousness.
* Current alcohol consumption exceeds 14 drinks per week.
* Self-reported illicit drug use.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Everyday Memory Questionnaire Revised | Day 24, Day 46, Day 77
  The Everyday Memory Questionnaire Revised (Royle & Lincoln, 2008) consists of 13 items that describe everyday events that might involve forgetting. Participants are asked how often on average they think each one has happened to them over the past month on a 5-point scale (0-4) and the total score is calculated as the sum of all responses. The minimum total score is 0 and the maximum is 52, with higher scores indicative of greater presence of memory difficulties. The outcome measure is the change in total score at the point of measurement compared to baseline at Day 1.
Change in General Cognitive Ability Composite Score | Day 77
  A composite score will be generated by taking the average of standardized outcome measures on tasks in the Standard Older Adult Cognitive Battery (SOACB), which consists of word list learning, complex figure copy, object naming, trail making, a vocabulary task, and matrix reasoning. The outcome measure is the change in the composite score reached on the task compared to baseline at Day 1.

SECONDARY OUTCOMES:
Change in Inhibitory Control Composite Score | Day 24, Day 46, Day 78
  The score is the mean of standardized dependent variables on tablet-based inhibitory control tasks. The outcome measure is the change in the composite score at the point of measurement compared to baseline at Day 2.
Training Experience Enjoyment | Day 24, Day 46
  Scores range from 1 to 5, with higher scores indicative of greater enjoyment of the training task enjoyment, subjective progress, and satisfaction of the training task
Training Experience Subjective Progress | Day 24, Day 46
  Scores range from 1 to 5, with higher scores indicative of greater subjective of the training task progress.
Training Experience Satisfaction Scale | Day 24, Day 46
  Scores range from 1 to 5, with higher scores indicative of greater satisfaction of the training task.
Training Experience Difficulty Scale | Day 24, Day 46
  Scores range from 1 to 10, with scores 1-3 indicating that the training was too easy, scores 4-7 indicating that the training was of appropriate difficulty, and scores 8-10 indicating that it was too difficult.
Exit Survey | Time Frame: Day 79
  Participants are asked 5 open-ended questions about their subjective experience of participating in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Jaeggi, PhD, Principal Investigator — Northeastern University; Aaron Seitz, Principal Investigator — Northeastern University
Locations (1):
- Northeastern University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Intervention materials and individual participant data (anonymized)
Supporting Information: Study Protocol
Time Frame: Data will be available persistently at the conclusion of the study.
Access Criteria: There are no access criteria